CLINICAL TRIAL: NCT05218278
Title: Dynamics of Light Chain of NFL as a Predictor Factor of Neurological Outcome in Patients With Out of Hospital Cardiac Arrest
Brief Title: NFL Dynamics as a Predictor Factor in Patients With Out of Hospital Cardiac Arrest
Status: Recruiting | Type: Observational
Sponsor: University Medical Centre Maribor (Other)
Responsible Party: Principal Investigator, Matej Strnad, Associate Proffessor, University Medical Centre Maribor
Other Study IDs: IRP-2021/01-01
Record Dates: First submitted 2022-01-17; First posted 2022-02-01 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Neurological Injury
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Trauma, Nervous System

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with favorable neurlogical outcome: CPC 1/2
- Patients with non-favorable neurological outcome: CPC3-5

SUMMARY:
To investigate the pharmacodynamics of light chain of NFL in patients with out-of hospital cardiac arrest after successful resuscitation and determine the difference in the serum levels of NFL in patients with favorable neurological outcome compared to those with non-favorable neurological outcome.

DETAILED DESCRIPTION:
To investigate the serum levels of the light chain of NFL at different time points after ICU admission (12, 24, 30, 36, 42, 48 hours after ICU admission) patients with out-of hospital cardiac arrest after successful resuscitation and determine the difference in the serum levels of NFL in patients with favorable neurological outcome compared to those with non-favorable neurological outcome.

ELIGIBILITY:
Inclusion Criteria:

* out-of-hospital cardiac arrest successfully resuscitated and admitted to the ICU

Exclusion Criteria:

* trauma, drowning, electrocution, less than 18 years of age,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-traumatic out-of-hospital cardiac arrest successfully resuscitated and admitted to the ICU.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The difference in the dynamics of serum NFL levels measurements in patients with favorable neurological outcome compared to patients with non-favorable neurological outcome | 3 years
  NFL levels

CONTACTS AND LOCATIONS:
Overall Officials: Matej Strnad, MD, PhD, Principal Investigator — University medical cenetr Maribor
Locations (1):
- University medical center Maribor, Maribor, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided
IPD that underlie results in a publication